CLINICAL TRIAL: NCT07094100
Title: Clinical Study of Cartilage Constructed by Autologous Bone Marrow Mesenchymal Stem Cells in Repairing Articular Cartilage Defects
Brief Title: Tissue Engineered Cartilage to Repairing Articular Cartilage Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TECOA-2021
Record Dates: First submitted 2025-06-25; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cartilage Injury; OA Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tissue-engineered cartilage to repair articular cartilage defects (Experimental)
  Interventions: Device: Tissue engineered cartilage

INTERVENTIONS:
Device: Tissue engineered cartilage — Cartilage constructed by autologous bone marrow mesenchymal stem cells

SUMMARY:
The joint cartilage constructed by combining bone marrow mesenchymal stem cells with three-dimensional materials has achieved the goal of repairing joint cartilage.

DETAILED DESCRIPTION:
Trauma, degeneration, inflammation, tumors, etc. can all cause damage to the cartilage of human joints. The cartilage has an extremely low self-repairing ability. Once damaged, the damage will become more and more severe over time, accelerating the occurrence and development of osteoarthritis, and causing varying degrees of joint dysfunction and reduced quality of life. Currently, traditional surgical treatments such as joint debridement, microfracture, and mosaic cartilage transplantation only apply to small-scale cartilage injuries, and long-term follow-up has found that the results are not satisfactory. The breakthrough in the core technology of in vitro constructing living cartilage based on tissue engineering principles has brought new hope for the physiological function reconstruction of joint cartilage damage. Cartilage was the first tissue to successfully regenerate using tissue engineering technology, but due to the limitation of the source of seed cells, no significant clinical breakthrough has been achieved. Studies have shown that bone marrow mesenchymal stem cells (BMSCs) are a type of cell with multi-directional differentiation potential (including cartilage and bone differentiation potential). Due to the fact that BMSCs can be autologously collected, the trauma is minimal, and the in vitro expansion ability is strong, therefore, they can meet the dual requirements of "quality and quantity" of seed cells for tissue engineering cartilage, and are very suitable for clinical application in the field of joint cartilage repair. More importantly, BMSCs have good cartilage formation ability. Our research group has established and invented a series of key technologies and methods for inducing BMSCs to form cartilage in vivo and in vitro in previous studies, and by applying BMSCs combined with three-dimensional degradable scaffold materials, we have been able to construct cartilage with a certain volume and morphology even biological joint tissues in vitro. At the same time, the application of autologous BMSCs for in vitro regeneration of cartilage has successfully repaired joint cartilage and bone composite defects in large animals, and especially has successfully carried out the exploratory clinical research of "in vitro construction of cartilage using autologous bone marrow mesenchymal stem cells for repairing joint cartilage defects", and after a 5-year follow-up, it has been confirmed that this technology can achieve satisfactory clinical repair effects. The research purpose of this application project is to use BMSCs combined with three-dimensional materials to construct joint cartilage to achieve the goal of repairing joint cartilage.

ELIGIBILITY:
Inclusion Criteria:

1. The patients' age ranges from 18 to 65 years old, and gender is not restricted;
2. The imaging results show that the epiphyseal growth is mature;
3. The defects or localized injuries of joint cartilage caused by trauma or other reasons;
4. The injured area is the distal weight-bearing surface of the femoral condyle of the knee joint, with no more than 4 lesions, and there is no injury to the cruciate ligaments;
5. The patients voluntarily sign and provide a written informed consent form and are willing to closely cooperate with the doctor's strict postoperative rehabilitation program.

Exclusion Criteria:

1. The patient is extremely overweight, with a body mass index greater than 35;
2. The lower limb alignment is valgus by more than 10° and varus by more than 5°;
3. Multiple ligament injuries;
4. There are numerous bad habits such as heavy smoking, drug abuse, and excessive alcohol consumption;
5. Has undergone open knee joint surgery within the past six months;
6. Has severe joint stiffness or fibrosis;
7. Has an allergic constitution or a history of allergic reactions to collagen;
8. Has mental abnormalities;
9. Cannot or is unwilling to undergo rehabilitation training;
10. Has primary cardiovascular diseases, lung diseases, endocrine and metabolic disorders, or other serious diseases that affect their daily life, such as tumors or AIDS;
11. Pregnant or lactating women, or those planning to conceive during the trial period;
12. Other acute or chronic diseases, for which the researchers consider surgery to be inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
KSS score | before the operation, at 3, 6, 12 and 24 months after the operation.
  subjective knee clinical and functional score (0-100)score.100 is better in function

SECONDARY OUTCOMES:
Koos scores | before the operation, at 3, 6, 12 and 24 months after the operation.
  subjective knee functional score (0-100)score.100 is better in function
Lysholm score | before the operation, at 3, 6, 12 and 24 months after the operation.
  subjective knee functional score (0-100)score.100 is better in function
WOMAC score | before the operation, at 3, 6, 12 and 24 months after the operation.
  The higher the index, the more severe the osteoarthritis. It is less than 80 for mild cases, 80 to 120 for moderate cases, and more than 120 for severe cases.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China